CLINICAL TRIAL: NCT00920868
Title: A Phase I Study of Capecitabine, Oxaliplatin, Bevacizumab, and Dasatinib for Patients With Advanced Solid Tumors With Expanded Cohort of Patients With Previously Untreated Metastatic Colorectal Cancer.
Brief Title: XAD - Xelox (Capecitabine + Oxaliplatin) + Bevacizumab + Dasatinib
Acronym: XAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herbert Hurwitz, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Herbert Hurwitz, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00010354
Record Dates: First submitted 2009-06-10; First posted 2009-06-15 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Solid Tumor; Metastatic Colorectal Cancer
Keywords: Phase I; Solid Tumor; Colorectal; Dasatinib; Sprycel; Bevacizumab; Avastin; Oxaliplatin; Eloxatin; Capecitabine; Xeloda; Duke; Any Solid Tumor (Phase I); Metastatic Colorectal Cancer (Expanded Cohort)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Dasatinib; Bevacizumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib 50mg (Experimental): Cohort 1
  Interventions: Drug: dasatinib; Drug: bevacizumab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: dasatinib — dasatinib at 50 mg PO BID)
  Other Names: Sprycel
Drug: bevacizumab — 7.5 mg/kg IV day 1
  Other Names: Avastin
Drug: Oxaliplatin — 130 mg/m2 IV day 1
  Other Names: Eloxatin
Drug: Capecitabine — 850 mg/m2 PO BID on days 1-14
  Other Names: Xeloda

SUMMARY:
The primary purpose of this study is to find the highest tolerated dose of the study drugs: capecitabine, oxaliplatin, bevacizumab, and dasatinib given in combination to subjects with advanced solid tumors. This will occur in the first part of the study (Phase I). Once this dose has been determined, it will be given to subjects with advanced metastatic colorectal cancer in the second part of the study (Phase II).

By giving these drugs in combination, researchers hope to evaluate the side effects of the study drugs in both groups, and to determine if this combination could possibly decrease or stabilize the cancer being treated.

Subjects will be enrolled at Duke University Medical Center (DUMC) and Rocky Mountain Cancer Center.

After satisfying eligibility and screening criteria, patients will be treated on 21 day cycles.

ABOUT THE STUDY DRUGS

* Capecitabine (Xeloda™) is an oral (taken by mouth) chemotherapy drug in tablet form made by Roche Laboratories Inc. Capecitabine has been approved for use by the Food and Drug Administration (FDA) for first line treatment (treatment that should be used for cancer that has not been treated yet) of metastatic colorectal cancer and also for metastatic breast cancer.
* Oxaliplatin (Eloxatin™) is an intravenous (given by injection into a vein) chemotherapy drug made by Sanofi-Synthélabo. This drug is also approved by the FDA for use in metastatic colorectal cancer.
* Bevacizumab (Avastin™) is a type of intravenous cancer treatment called anti-angiogenic therapy (a type of therapy to treat cancer that interferes with blood flow to the tumor, thereby stopping tumor growth, and possibly leading to tumor shrinkage) made by Genentech Inc. Bevacizumab is approved by the FDA for first line treatment of metastatic colorectal cancer in combination with other chemotherapy.
* Dasatinib (Sprycel™) is an oral drug made by Bristol Myers Squib, Inc (BMS). Dasatinib is approved by the FDA for the treatment of chronic myeloid leukemia (CML), acute lymphoblastic leukemia or for patients that are resistant to a medicine called imatinib mesylate (Gleevec™ ).

ELIGIBILITY:
Inclusion Criteria:

Criteria Specific for Dose Escalation (Phase I)

1. Patients must have histologically confirmed solid tumor malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective, or for whom capecitabine, oxaliplatin, and/or bevacizumab would be considered a standard therapy or therapeutic option.
2. Patients must not have had radiation therapy, hormonal therapy, biologic therapy or chemotherapy for cancer within the 28 days prior to study day 1.

Criteria Specific for Expanded Cohort Portion of Trial Only

1. Histologically documented adenocarcinoma of the colon or rectum that is metastatic/recurrent disease
2. No prior chemotherapy for metastatic/recurrent colorectal cancer. Patients may have received a radiosensitizing dose of 5-fluorouracil or capecitabine for the treatment of local disease in the localized or metastatic setting.
3. No history of other carcinomas within the last five years, except cured non-melanoma skin cancer, curatively treated in-situ cervical cancer, or localized prostate cancer
4. Disease must be measurable by Response Evaluation Criteria In Solid Tumors (RECIST) criteria

Inclusion Criteria for All Participants

1. Age >18 years.
2. Karnofsky performance status > 70%.
3. Life expectancy of at least 3 months.
4. Patients must have adequate organ and marrow function as defined below:
5. Sexually active women of childbearing potential must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized.
6. All women of child bearing potential (WOCBP) MUST have a negative pregnancy test within 7 days prior to first receiving investigational product.
7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria for ALL Subjects:

1. Patients who have had radiation therapy, hormonal therapy, biologic therapy, or chemotherapy for cancer within the 28 days prior to day 1 of the study (ie - first day of study drug treatment).
2. Patients who have received any other investigational agents within the 28 days prior to day 1 of study drug treatment.
3. Patients with known central nervous system (CNS) metastases.
4. Inadequately controlled hypertension
5. Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
6. Symptomatic peripheral vascular disease
7. Evidence of bleeding diathesis or coagulopathy. Patients on full-dose anticoagulation are permitted to enroll provided that they have been clinically stable on anti- coagulation.
8. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1 of study drug treatment
9. Core biopsy or other minor surgical procedure excluding placement of a vascular access device, within 7 days prior to expected start of treatment.
10. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study day 1
11. Serious, non-healing wound, ulcer, or bone fracture
12. Proteinuria at screening
13. Any prior history of hypertensive crisis or hypertensive encephalopathy
14. New York Heart Association (NYHA) Grade II or greater congestive heart failure
15. History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 6 months prior to study treatment day 1
16. History of stroke or transient ischemic attack within 6 months prior to study treatment day 1
17. History of intolerance or hypersensitivity to prior treatment with capecitabine, oxaliplatin, bevacizumab and/or dasatinib.
18. No previous treatment with dasatinib.
19. Prior unanticipated severe reaction to fluoropyrimidine therapy, or known hypersensitivity to 5-fluorouracil, or known dihydropyrimidine dehydrogenase (DPD) deficiency.
20. Patient with grade 2 or greater peripheral neuropathy
21. Chronic treatment with systemic steroids or another immunosuppressive agent.
22. Other concurrent severe and/or poorly controlled medical condition that could compromise safety of treatment as so judged by treating physician.
23. A known history of HIV seropositivity,hepatitis C virus, acute or chronic active hepatitis B infection, or other serious chronic infection requiring ongoing treatment.
24. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter drug absorption (e.g., inflammatory bowel disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or significant small bowel resection)
25. Patients unwilling to or unable to comply with the protocol
26. Diagnosed or congenital long QT syndrome
27. Any history of clinically significant ventricular arrhythmias
28. Prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (> 450 msec)
29. Pleural effusion grade > 2.
30. Patients currently taking drugs that are generally accepted to have a risk of causing Torsades de Pointes including:
31. History of significant bleeding disorder unrelated to cancer
32. Patients actively taking proton pump inhibitors or H2 antagonists will be excluded from this study.
33. Any psychiatric illness/social situations that would limit safety or compliance with study requirements
34. Medications that inhibit platelet function (except low dose aspirin as defined in study protocol)
35. Use of medications that are either Cytochrome P450 3A4 (CYP3A4) inhibitors or inducers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose(MTD)/recommended phase II dose (RPTD) of capecitabine/oxaliplatin/bevacizumab/dasatinib for patients with advanced solid tumors. | 9 months

SECONDARY OUTCOMES:
To further describe dose-limiting and non-dose-limiting toxicities associated with this regimen. | 12 months
To describe clinical activity (partial response (PR), complete response (CR) or stable disease (SD)>6 months, time to progression, and overall survival) associated with this regimen for patients with previously untreated metastatic and/or re | 2 years
To explore any correlation between blood, urine, and paraffin biomarkers and clinical outcomes | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Herbert I Hurwitz, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Duke Univeristy Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Strickler JH, McCall S, Nixon AB, Brady JC, Pang H, Rushing C, Cohn A, Starodub A, Arrowood C, Haley S, Meadows KL, Morse MA, Uronis HE, Blobe GC, Hsu SD, Zafar SY, Hurwitz HI. Phase I study of dasatinib in combination with capecitabine, oxaliplatin and bevacizumab followed by an expanded cohort in previously untreated metastatic colorectal cancer. Invest New Drugs. 2014 Apr;32(2):330-9. doi: 10.1007/s10637-013-0042-9. Epub 2013 Nov 1. PMID 24173967